CLINICAL TRIAL: NCT01457378
Title: Assessment of Gastrointestinal Symptoms and Health-related Quality of Life in Healthy People and Patients With Irritable Bowel Syndrome
Brief Title: Gastrointestinal Symptoms in Healthy Subjects and Patients With Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Other Study IDs: NU357
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Gastrointestinal symptoms; healthy subjects; IBS; HRQoL; questionnaires
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers: 100 healthy volunteers
- IBS Subjects: 100 IBS Subjects

SUMMARY:
The aim of this study performed in Irritable Bowel Syndrome (IBS) subjects and healthy patients is to demonstrate the ability of composite score of frequency of gastrointestinal symptoms to discriminate healthy subjects and IBS patients. The properties of this questionnaire of composite score of gastrointestinal symptoms frequency will be compared to other validated questionnaires (severity of IBS symptoms and HRQoL).

ELIGIBILITY:
Inclusion Criteria:

* for Healthy subjects :
* Healthy women and men free-living subject aged from 18 to 65 years.
* Subject with a body mass index between 18 and 30, bounds included.
* Subject having given written consent to take part in the study.
* Chronic medical treatment-free excluding contraceptive and stable Hormonal Replacement Therapy
* for IBS Patients :
* IBS women and men free-living subject aged from 18 to 65 years
* Subject with a diagnosis of IBS according to Rome III criteria: recurrent abdominal pain or discomfort at least 3 days per month in the last 3 months associated with 2 or more of the following: improvement with defecation; onset associated with a change in frequency of stool; onset associated with a change in form (appearance) of stool.
* Subject with a diagnosis of IBS according to Rome III criteria with symptom onset at least 6 months prior to diagnosis.
* Subject having an IBS-SSS score higher or equal to 75 corresponding to an active phase of IBS symptoms.
* Subject having given written consent to take part in the study.

Exclusion Criteria:

* for Healthy subjects :
* Subject who, in the past, has consulted a general practitioner or a gastroenterologist for (IBS) or any other functional bowel disease including constipation and diarrhoea.
* Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease
* Subject treated with any chronic medical treatment that, in the investigator's opinion could interfere with the GI tract.
* Subject who underwent general anaesthesia in the preceding 4 weeks.
* Pregnant subject or breast-feeding subject at the time of the study.
* Subject with known immunosuppression
* Subject with any known food allergy
* Subject involved in any other clinical study within the preceding month or in exclusion period after another clinical study.
* Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.
* Subject not able to read, to understand and/or to answer to the questionnaires.
* for IBS Patients :
* If a subject fulfils with one of the following criteria, he/she must be excluded from the study:
* Subject with a diagnosis of IBS with clinical signs of alarm (rectorragy, fever, associated inflammatory articular signs, recent weight loss).
* Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease.
* Subject who underwent general anaesthesia in the preceding 4 weeks.
* Pregnant subject or breast-feeding subject at the time of the study.
* Subject involved in any other clinical study within the preceding month or in exclusion period after another clinical study.
* Taking antidepressant or analgesic drugs.
* Subject not able to read, to understand and/or to answer to the questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy subjects and adult IBS patients (Rome III criteria, all subtype)
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Eurofins Optimed, Gières
  - Biofortis, Nantes

REFERENCES:
- [Derived] Azpiroz F, Guyonnet D, Donazzolo Y, Gendre D, Tanguy J, Guarner F. Digestive Symptoms in Healthy People and Subjects With Irritable Bowel Syndrome: Validation of Symptom Frequency Questionnaire. J Clin Gastroenterol. 2015 Aug;49(7):e64-70. doi: 10.1097/MCG.0000000000000178. PMID 25014236